CLINICAL TRIAL: NCT02007694
Title: Noradrenergic Manipulation and Virtual Reality Exposure Therapy in Phobic Participants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Paul M.G.Emmelkamp, Prof. dr., VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-KP-2464
Record Dates: First submitted 2013-03-20; First posted 2013-12-11 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Phobic Disorders
Keywords: Phobic Disorders (Fear of Flying and acrophobia); Virtual Reality Exposure Therapy; Fear extinction; propranolol; Yohimbine
MeSH Terms: conditions — Phobic Disorders; Aerophobia; Acrophobia | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- VRET plus Yohimbine (Active Comparator): Virtual Reality Exposure Therapy combined with the administration of yohimbine.
  Interventions: Behavioral: Virtual Reality Exposure Therapy (VRET)
- VRET plus propranolol (Active Comparator): Virtual Reality Exposure Therapy combined with the administration of propranolol
  Interventions: Behavioral: Virtual Reality Exposure Therapy (VRET)
- VRET plus placebo (Placebo Comparator): Virtual Reality Exposure Therapy combined with the administration of a non-active placebo pill
  Interventions: Behavioral: Virtual Reality Exposure Therapy (VRET)

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy (VRET) — Graded exposure to feared specific stimulus by computer-generated 3D virtual environments.

SUMMARY:
Recent advances in animal research have identified pharmacological agents that appear to both accelerate and consolidate extinction learning. One cognitive enhancers is Yohimbine hydrochloride (YOH). A finding in animal literature is that the administration of YOH during extinction trials accelerates fear reduction and may convert ineffective exposures in to successful ones. It is thought that the mechanism of enhanced emotional memory is through elevated norepinephrine. However, recent findings demonstrate mixed results. In a randomized controlled trial claustrophobic participants underwent exposure in combination with YOH or placebo. The YOH group showed significantly better results on anxiety improvement than the placebo group. In a more recent study with participants with fear of flying no additional benefits of YOH were demonstrated. Therefore, we intend to replicate and extend these studies by enhancing the dose of YOH in combination with VRET and by extending our experimental design with another group which receives propranolol in combination with VRET. Propranolol is β-adrenergic receptor antagonist, which has proven to disrupt reconsolidation in healthy humans. In this randomized controlled trial a between groups design is chosen to further characterize the differential within and between trial extinction and to enhance possible between groups effects. Sixty participants with fear of flying or fear of heights will be randomly assigned to one of the following three conditions 1) VRET plus YOH, 2) VRET plus Propranolol, or 3) VRET plus placebo. Participants in all conditions will be offered three sessions of VRET over a period of two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Marked fear of flying or acrophobia, indicated by a subjective fear rating of moderate or higher on anxiety specific measures.

Being older than 18 years and younger than 75 years.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
FAS (Flight Anxiety Situations Questionnaire) | Pre- (baseline) and post-assessment (after treatment termination, within 3 weeks after first treatment session) and 3 month follow up (3 month after post assessment)
  The FAS is 32-item, self-report inventory designed to measure anxiety related to flying experienced in different situations. The FAS is divided into three subscales: the Anticipation scale, which represents situations before the actual flight, the In-flight scale, which refers to situations during a flight and the Generalized flight scale.
AQ (Acrophobia Questionnaire) | Pre- (baseline) and post-assessment (after treatment termination, within 3 weeks after first treatment session) and 3 month follow up (3 month after post assessment)
  The AQ (Cohen, 1977) is a 40-item self-report measure to assess anxiety in height situations. The AQ measures anxiety and avoidance behavior relative to height situations. Subject can express their fear on a scale ranging from 0-6, whereby 0 stands for "no fear at all" and 6 for "almost panic" (ranging from 0-120).
WAQ (Weekly Anxiety Questionnaire) | In session 1, 2 and 3 and Pre- (baseline) and post-assessment (after treatment termination, within 3 weeks after first treatment session) and 3 month follow up (3 month after post assessment)
  The WAQ is an author-constructed transdiagnostic anxiety questionnaire to rate severity of experienced general anxiety. The WAQ is a 10-item self-report measure on which participants can rate their experienced anxieties. Ratings can be scored on a five-point Likert scale ranging from "not at all" to "permanently".

SECONDARY OUTCOMES:
FAM (Flight Anxiety Modalities Questionnaire) | Pre- (baseline) and post-assessment (after treatment termination, within 3 weeks after first treatment session) and 3 month follow up (3 month after post assessment)
  The FAM is 23-item, self-report inventory designed to measure how fear of flying can be expressed. On a five-point-likert scale the intensity of fear can be rated. The FAM is divided into two subscales: the Somatic Modality, which represents the physical symptoms and the Cognitive Modality, which measures distressing cognitions.
ATHQ (Attitude towards heights questionnaire) | Pre- (baseline) and post-assessment (after treatment termination, within 3 weeks after first treatment session) and 3 month follow up (3 month after post assessment)
  The ATHQ contains six questions assessing the attitude towards heights (range 0-60).
DASS (Depression Anxiety Stress Scale) | Pre- (baseline) and post-assessment (after treatment termination, within 3 weeks after first treatment session) and 3 month follow up (3 month after post assessment)
  The DASS is 42-item self-report measure that assesses level of depression, anxiety, and stress over the previous week. Each scale consists of 14 items, which are grouped into smaller subscales. The depression scale consists of the following subscales: dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia and inertia. The anxiety scale consists of: autonomic arousal, skeletal musculature effects, situational anxiety and subjective experience of anxious affect. The stress scale consists of: difficulty relaxing, nervous arousal, easily agitated, irritable/overreactive and impatient. The internal consistency of the DASs is good to excellent (Cronbach's alpha ranging from .88 to .96; Brown et al., 1997).
PIT (Prospective Imagery Task) | Pre- (baseline) and post-assessment (after treatment termination, within 3 weeks after first treatment session) and 3 month follow up (3 month after post assessment)
  The PIT is based on MacLeod and Byrne, (1996) and Stöber, (2000) and will be used to measure imagery for 10 positive and 10 negative prospective events. As in Holmes, Lang, et al. (2008), subjects will be asked to rate the vividness of prospective positive events (e.g., "You will have lots of energy and enthusiasm") or negative events (e.g., "Someone close to you will reject you") on a 5-point scale (1 = no image at all; 5 = very vivid).
ASI (Anxiety Sensitivity Inventory) | Pre- (baseline) and post-assessment (after treatment termination, within 3 weeks after first treatment session) and 3 month follow up (3 month after post assessment)
  The ASI is a 16-items self-report questionnaire, measuring fear of anxiety-related symptoms. Each item is rated on a five-point likert scale ranging from 0 (very little) to 4 (very much). The ASI is scored by summing all items; possible scores range from 0 to 64, with higher scores reflecting higher levels of anxiety sensitivity.
SUDs (Subjective Units of Discomfort) | Every 3 minutes during exposure (exposure will be done twicely 25 minutes every therapy session. Thus, starting at minute 1 every 3 minute a SUD will be asked. After a break of 10 minutes, exposure will start again (25 minutes).
  Subjective Units of Discomfort (SUDs) will be taken every 3 minutes to monitor patients' subjective anxiety (Wolpe, 1990).

OTHER OUTCOMES:
QMI (Questionnaire upon Mental Imagery) | Pre-assessment (baseline); first treatment session will follow within 3 weeks
  The QMI measures vividness of imagery typically experienced by participants across seven sensory modalities: visual, auditory, cutaneous, gustatory, kinaesthetic, olfactory, and organic. The QMI is a reliable instrument containing 35 items. The items rate the vividness on a seven point scale (1 = "I perceive it perfectly clearly, as if it were real"; 7 = "I think about it, but I cannot imagine it").
IPQ (Igroup Presence Questionnaire) | Post session 1, 2 and 3 (all within 2 weeks, maximum 3 weeks)
  The IPQ is a 14-item, self-report inventory designed to measure to what degree participants experience the virtual environments as real.The IPQ consists of three underlying factors, which refer to respectively: 1) the spatial presence, meaning which is the sense of really being in a virtual environment, 2) involvement: the attention which is paid to the real world and to the virtual environments and 3) the realness of the virtual world, which refers to the reality jugdement of the virtual world. The subject can give an indication of how real the virtual world is on a scale ranging from -3 to +3, respectively "completely disagree" and "completely agree".
SSQ (Simulator Sickness Questionnaire) | Post session 1, 2 and 3 (all within 2 weeks with a maximum of 3 weeks)
  The SSQ is a 27-item self-report questionnaire designed to measure whether subjects experienced any physiological symptoms during and after being in the virtual environments. Participants can give an indication whether and to what degree they experienced twenty-seven physiological symptoms: with underlying factors tiredness, anxiety or panic and traumatic memory.
EEQ (Exposure Experience Questionnaire) | Post session 1, 2 and 3 (all within 2 weeks with a maximum of 3 weeks)
  The EEQ is a 7-item author-constructed self-report questionnaire we designed to measure the degree of anxiety and presence after virtual reality exposure therapy.
TGAQ (Treatment Gain and Attribution Questionnaire) | Post-assessment (inmediately after the last treatment session)
  The TGAQ is based on the TGAQ from Powers and colleague's and (Powers et al., 2008) is a fourteen-item scale assesses participants' perceptions of their level of improvement and the extent to which the herbal supplement facilitated or interfered with their exposure treatment. The four dimensions are rated using 100-point visual analogue scales, including the following: (a) overall improvement (not at all improved to much improved), (b) medication interference (not at all detrimental to extremely detrimental), (c) medication facilitation (not at all helpful to extremely helpful), and (d) exposure facilitation (not at all helpful to extremely helpful).
Drug guess | Post-assessment (inmediately after the last treatment session)
  A questionnaire consisting of 5 questions concerning the medication and its possible effects will be used to assess whether participants are aware in which drug condition they participate. Participants are asked whether they had received YOH/propranolol or placebo and rated on a scale ranging from 0 (not sure at all) to 100 (definite) how sure they were that their guess was right.
Self-efficacy questionnaire | Pre- and post session 1, 2 and 3 (all within 2 weeks with a maximum of 3 weeks)
  The self-efficacy questionnaire is a self-report inventory designed to measure the degree of self-efficacy subjects experienced with respect to the phobic situation. The inventory consists of five items on self-efficacy in phobic situations. The items represent five different themes 1) the capability to reduce the experienced fear, 2) to think clearly, 3) to control for ones own actions, 4) to control anxious thoughts and feelings and 5) to stay in the situation while experiencing intense fear. The participant can give an indication by giving a percentage representing their evaluation of their own capability.
Cognitions Questionnaire | Post session 1, 2 and 3 (all within 2 weeks with a maximum of 3 weeks)
  The cognition questionnaire is a self-report inventory designed to investigate the level of positive and negative cognitions subjects have about themselves. The questionnaire consists of 30 items for fear of flying which can be scored on a five-point Likert scale ranging from "not at all" to "permanently".
Expectancy | Pre-assessment (baseline); first treatment session will follow within 3 weeks
  Participants expectancy about the outcome will be rated on a 5-item self-report scale based on the Borkovec and Nau (1972) expectancy of improvement scale (0%-100%).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Emmelkamp, PhD, Principal Investigator — University of Amsterdam
Locations (1):
- University of Amsterdam, Amsterdam, North Holland, Netherlands